CLINICAL TRIAL: NCT02906033
Title: The Effect of A New Perioperative Practice Model on Patient, Nursing And Organisational Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital District of Helsinki and Uusimaa (Other)
Collaborators: University of Turku (Other); Karlstad University (Other)
Responsible Party: Principal Investigator, Kristiina Junttila, Director of Nursing Research Center, Hospital District of Helsinki and Uusimaa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: TYH2014211; U1111-1185-9612 (Other: WHO: The Universal Trial Number (UTN))
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Results first posted 2021-12-06 (Actual); Last update posted 2021-12-06 (Actual); Status verified 2021-10

CONDITIONS: Arthroplasties, Hip Replacement; Arthroplasties, Knee Replacement
Keywords: Surgical Procedures, Operative; Operating Rooms; Quality of Life; Surgery-related anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): New perioperative practice model.
  Interventions: Other: New perioperative practice model
- Control group (No Intervention): Traditional practice model.

INTERVENTIONS:
Other: New perioperative practice model — The one and same anesthesia nurse takes care of the patient during the entire perioperative process and even pays the patient a visit to the ward the day after surgery.
  Arms: Intervention group

SUMMARY:
The aim of the study is to improve the surgical patients' care process. The objective is to explore the effect of a new perioperative practice model on 1) patient outcomes (satisfaction, surgery-related anxiety and quality of life), 2) nursing outcomes (organizational engagement), and 3) organization outcomes (timeline of surgical care process).

DETAILED DESCRIPTION:
Study design:

A longitudinal untreated control group design with pre- and posttests will be followed.

Setting and sampling:

The study will be conducted at the Helsinki University Hospital; more specifically at the operating department K of the Peijas Hospital. The randomized patient sampling will include voluntary adult surgical patients undergoing a hip or a knee replacement procedure. The patients will be recruited during their preoperative visit (approx. 2-3 weeks prior to the operation), and an informed consent will be obtained. Approximately 12-16 patients per day are scheduled for the preoperative visits, summing up to 60-80 recruitments per week. A control group (Group A) and an experimental (intervention) group (Group B) will be formed. The sample size was checked with power analysis (2 sided test) with the following parameters: value for α = 0.05, value for power 0.8, and value for common standard deviation 0.1. The sample size for both groups (A and B) was set at 175. Considering the potential drop-out, approx. 30%, the final sample size was determined to be 245 per group. The randomization will be performed by an independent third party (i.e., nurses at the preoperative clinic). The eligible patients will draw one of two cards; one indicating that an invitation to participate the study will be given to them, and the other being empty. Patients for the Group A will be recruited on the first week and the patients for the Group B on the second week. This pattern will be repeated until the desired amount of patients is recruited. This stratification will ensure that the two groups will not be contaminated in the ward where the post-operative visits will be carried out.

Data collection and instruments:

The patient data will be collected with 1) The Good Perioperative Nursing Care Scale developed by Leinonen and Leino-Kilpi (2001); 2) 15D; a generic, 15-dimensional, self-administered instrument for measuring health related quality of life among adults, developed by professor Sintonen; and 3) STAI, The State-Trait Anxiety Inventory; a definitive instrument for measuring anxiety in adults developed by Dr. Spielberger. The following demographic data from the participants will be collected: age, gender, diagnosis, procedure, and ASA-classification.

Intervention:

Traditionally during the intra- and postoperative phases of surgical care, the patient is cared for by several nurses; i.e. by an anesthetic nurse in the operating room and by a recovery room nurse in the Post Anesthesia Care Unit (PACU). Furthermore, the pre- and postoperative visits to the surgical patients are rare in Finland; mainly due to resources and new surgical processes where patients arrive to the hospital in the morning of the scheduled procedure.

Basically, the new perioperative practice model denotes that the one and same nurse will meet the patient at his/her arrival to the operating department, and will care for the patient both in the operating room and in the PACU. Thus, the nursing care in the operating room and in the PACU remains the same, but will be organized in a new way which focuses on the patient centered individual care and the continuity of care. Furthermore, the same nurse will visit the patient at the surgical unit on the first postoperative day.

A uniform content for the postoperative visits will be defined to ensure consistency of the intervention. The nurse will ask the patients if they have any questions or concerns regarding the procedure, how they have experienced their perioperative care, what they very satisfied with and what they would have desired to be different or would expect in the future from their care. The main aim of the visits is to meet the patient as an individual with individual needs and desires.

According to the previous research results this new way to allocate personnel did not cause additional resource needs and did not in any way harm the care of other patients who did not participate in the study.

Data analysis:

Descriptive, inferential and advanced statistical analyses will be used.

ELIGIBILITY:
Inclusion Criteria:

* the patient has been scheduled for a primary elective hip or a knee replacement procedure under spinal anesthesia
* the patient is 18 years of age or older
* the patient is able to participate in the study either in Finnish or Swedish
* the patient is able to give his/her written consent to participate the study
* the patient is willing to participate the study
* the patients operation time is scheduled on Monday through Thursday in the operating department K in the Peijas hospital

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristiina Junttila, PhD, Study Director — Hospital District of Helsinki and Uusimaa
Locations (1):
- Peijas Hospital / Helsinki University Hospital, Vantaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pulkkinen M, Jousela I, Sintonen H, Engblom J, Salantera S, Junttila K. A randomized clinical trial of a new perioperative practice model on anxiety and health-related quality of life in arthroplasty patients. Nurs Open. 2021 Jul;8(4):1593-1605. doi: 10.1002/nop2.776. Epub 2021 Feb 12. PMID 33576579
- [Derived] Pulkkinen M, Jousela I, Engblom J, Salantera S, Junttila K. The effect of a new perioperative practice model on length of hospital stay and on the surgical care process in patients undergoing hip and knee arthroplasty under spinal anesthesia: a randomized clinical trial. BMC Nurs. 2020 Jul 31;19:73. doi: 10.1186/s12912-020-00465-3. eCollection 2020. PMID 32765189

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Excluded due to general anesthesia: N=64
Period: Baseline
Arm/Group | Intervention Group | Control Group
Started | 231 | 222
15 D at Baseline (Analyzed at baseline for 15 D) | 211 | 189
STATE at Baseline (Analyzed at baseline for STATE anxiety) | 199 | 190
TRAIT at Baseline (Analyzed at baseline for TRAIT anxiety) | 194 | 189
Completed | 194 (Analyzed at baseline for 15 D and STATE anxiety and TRAIT anxiety) | 189 (Analyzed at baseline for 15 D and STATE anxiety and TRAIT anxiety.)
Not Completed | 37 | 33
Not completed — Protocol Violation | 37 | 33
Period: Follow-up
Arm/Group | Intervention Group | Control Group
Started | 194 | 189
15 D at Follow-up (Analyzed for 15 D at follow-up) | 151 | 135
STATE at Follow-up (Analyzed for STATE anxiety at follow-up) | 154 | 135
TRAIT at Follow-up (Analyzed for TRAIT anxiety at follow-up) | 148 | 127
Completed | 148 (Analyzed for 15 D and STATE anxiety and TRAIT anxiety at follow-up) | 127 (Analyzed at follow-up 15 D and STATE anxiety and TRAIT anxiety.)
Not Completed | 46 | 62
Not completed — Lost to Follow-up | 46 | 62

BASELINE CHARACTERISTICS:
Population: In all, for the intervention group, 260 participants were enrolled. Of the, 231 received allocated intervention (n=29 excluded due to general anesthesia).
  For the control group, 257 participants were enrolled. Of them, 222 received standard perioperative care (n=35 excluded due to general anesthesia).
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 231 | 222 | 453
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Enrolled participants
  years | 67.0 (10.41) | 68.0 (10.48) | 67.0 (10.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 139 | 285
  Male | 85 | 83 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 231 | 222 | 453
Region of Enrollment [Number; unit: participants]
  Finland | 231 | 222 | 453

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Follow-up in Health Related Quality of Life
Description: The 15D is a generic, comprehensive, 15-dimensional, standardized, self-administered measure of health-related quality of life (HRQoL) that can be used both as a profile and single index score measure.
  The 15 dimensions are: mobility, vision, hearing, breathing, sleeping, eating, speech, excretion, usual activities, mental functioning, discomfort and symptoms, depression, distress, vitality, and sexual activity The respondent chooses one of the five levels for each dimension that best describes his or her state of health at present moment; the best level is 1 and the worst is 5.
  The single index score (15D score), representing the overall HRQoL on a 0-1 scale (1=full health, 0=being dead). The results in Outcome Measure Data Table describe the changes from baseline to follow-up within the intervention group and the control group.
Time Frame: Baseline and at 3 months follow up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 151 | 135
score on a scale | 0.059 [0.036 to 0.081] | 0.055 [0.031 to 0.078]

2. Secondary Outcome: Change in Surgery-related STATE Anxiety From Baseline to Follow-up
Description: The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes.
  This instrument is composed of STATE and TRAIT scales, each of which has twenty items. The STATE items evoke feelings on a 4-point Likert scale, with responses ranging from 1 (not at all) to 4 (very much). The TRAIT items evoke how the respondent feels in general on a frequency scale ranging from 1 (hardly ever) to 4 (almost always). The scores of both STATE and TRAIT scales range from 20 to 80 scores.
  According to the raw score, anxiety is classified as low (20-39), moderate (40-59) or high (60-80). The results in Outcome Measure Data Table describe the changes from baseline to follow-up within the intervention group and the control group.
Time Frame: Baseline and at 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 154 | 135
score on a scale | -4.91 [-8.02 to -1.79] | -5.21 [-8.47 to -1.95]

3. Secondary Outcome: Quality of Perioperative Care as Experienced by Surgical Patients
Description: Good Perioperative Nursing Care Scale is a constructed questionnaire which contains 36 statements measuring the quality of care, which are summarized into nine quality categories (sum variables/subscales): Pain management (n=5 statements), Temperature maintenance (n=2), Technical skills (n=4), Information (n=6), Encouragement (n= 3), Respect (n= 3), Staff characteristics (n= 5), Environment (n= 6) and Process (n= 2).
  The quality statements are answered with a five-point Likert scale (fully agree, 5 points - fully disagree, 1 point) with a neutral option "neither agree nor disagree" and an option "cannot evaluate this aspect". The value of each averaged sum variable/subscale varies from 1 to 5. In the analysis, the responses of "cannot evaluate this aspect" were excluded. The better the mean value is, the more positive experience the participant has of the quality of care.
Time Frame: One-point measurement on the day of discharge (on average on the 3rd day after surgery)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 219 | 217
score on a scale
  Sum variable "Pain management" | 4.85 [4.78 to 4.91] | 4.83 [4.76 to 4.89]
  Sum variable "Technical skills" | 4.95 [4.92 to 4.98] | 4.90 [4.84 to 4.95]
  Sum variable "Information" | 4.61 [4.47 to 4.74] | 4.58 [4.44 to 4.71]
  Sum variable "Encouragement" | 4.61 [4.49 to 4.72] | 4.56 [4.42 to 4.70]
  Sum variable "Respect" | 4.87 [4.80 to 4.94] | 4.76 [4.68 to 4.85]
  Sum variable "Staff characteristics" | 4.89 [4.84 to 4.94] | 4.83 [4.75 to 4.90]
  Sum variable "Environment" | 4.79 [4.71 to 4.87] | 4.81 [4.74 to 4.88]
  Sum variable "Temperature management" | 4.90 [4.84 to 4.96] | 4.95 [4.92 to 4.99]
  Sum variable "Process" | 4.71 [4.60 to 4.82] | 4.51 [4.35 to 4.68]

4. Secondary Outcome: Change in Surgery-related TRAIT Anxiety From Baseline to Follow-up
Description: The State-Trait Anxiety Inventory (STAI) is a commonly used measure of trait and state anxiety. It can be used in clinical settings to diagnose anxiety and to distinguish it from depressive syndromes.
  This instrument is composed of STATE and TRAIT scales, each of which has twenty items. The STATE items evoke feelings on a 4-point Likert scale, with responses ranging from 1 (not at all) to 4 (very much). The TRAIT items evoke how the respondent feels in general on a frequency scale ranging from 1 (hardly ever) to 4 (almost always). The scores from both STATE and TRAIT scales range from 20 to 80 scores.
  According to the raw score, anxiety is classified as low (20-39), moderate (40-59) or high (60-80). The results in Outcome Measure Data Table describe the changes from baseline to follow-up within the intervention group and the control group.
Time Frame: Baseline and at 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 148 | 127
score on a scale | -0.76 [-3.54 to 2.02] | -2.05 [-4.98 to 0.88]

ADVERSE EVENTS:
Time Frame: As an interventional nursing practice study, the adverse events were not anticipated nor collected.
Description: As an interventional nursing practice study, the adverse events were not anticipated nor collected.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT02906033/Prot_SAP_000.pdf